CLINICAL TRIAL: NCT03194048
Title: Effect of Functional Chewing Training on Tongue Thrust and Drooling in Children With Cerebral Palsy: A Randomised Controlled Trial
Brief Title: Effect of Functional Chewing Training on Tongue Thrust and Drooling in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İNAL, Özgü İNAL, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: özgü inal
Record Dates: First submitted 2017-06-13; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Mastication Disorder
Keywords: drooling; tongue thrust
MeSH Terms: conditions — Sialorrhea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Chewing Training (Experimental): Children with CP and have tongue thrust included this group.
  Interventions: Other: Functional Chewing Training
- Control (Active Comparator): Children with CP and have tongue thrust included this group.
  Interventions: Other: Classical Oral Motor Exercises

INTERVENTIONS:
Other: Functional Chewing Training — FuCT;
  * Family training
  * Providing optimal sitting posture for children to support oral sensorimotor functions
  * Positioning the food to the molar area during every meal to stimulate lateral and rotational tongue movements
  * Massage of the upper and lower gums through the front teeth to molar area
  * Chewing training to stimulate lateral and rotational tongue movements
  * Gradually increasing the food consistency, for 12 weeks in 5 sets (1 set = 20 min) each day
  Other Names: FuCT
  Arms: Functional Chewing Training
Other: Classical Oral Motor Exercises — Classical Oral Motor Exercises;
  * Family training
  * passive and active lip and tongue exercises, for 12 weeks in 5 sets (1 set = 20 min) each day
  Arms: Control

SUMMARY:
This study examined the effect of Functional Chewing Training(FuCT) on tongue thrust and drooling in children with cerebral palsy.

DETAILED DESCRIPTION:
Children were divided into two groups: The FuCT group and control group receiving classical oral motor exercises. Each group received training for 12 weeks. Oral motor assessment was performed. Chewing performance level was determined with the Karaduman Chewing Performance Scale(KCPS). Tongue thrust severity was evaluated with the Tongue Thrust Rating Scale(TTRS). The Drooling Severity and Frequency Scale(DSFS) was used to evaluate drooling severity and frequency. The evaluations were performed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with cerebral palsy
* aged between 4-6 years
* fed by orally
* had tongue thrust

Exclusion Criteria:

* children who were unable the sitting position

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2015-12-20 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Tongue Thrust Rating Scale | 12 weeks
  Tongue thrust for each child is scored while they are feeding.

SECONDARY OUTCOMES:
The Drooling Severity and Frequency Scale | 12 weeks
  Parents were asked how often and in which severity experiencing drooling their children.

CONTACTS AND LOCATIONS:
Overall Officials: Özgü İnal, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rempel GR, Colwell SO, Nelson RP. Growth in children with cerebral palsy fed via gastrostomy. Pediatrics. 1988;82:857-862. Allen MC, Capute A. The evolution of primitive reflexes in extremely premature infants. Pediatr Res. 1986;20:1284-1289. Blasco PA. Primitive reflexes: their contribution to the early detection of cerebral palsy. Clinical pediatrics. 1994;33:388-397. Singh S, Dua P, Jain S. Habit breaking appliance for tongue thrusting-a modification. Indian J Dent Sci. 2011;3:10.